CLINICAL TRIAL: NCT06313580
Title: Spices for Cultivating a Healthy Gut Microbiome and Cardiometabolic Profile: the SPICE Study
Brief Title: Spices for Cultivating a Healthy Gut Microbiome and Cardiometabolic Profile
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 22-1055
Record Dates: First submitted 2024-01-03; First posted 2024-03-15 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cardiometabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Yogurt

STUDY DESIGN:
Intervention Model Description: In a single blind crossover design, participants are randomized to 4 weeks of yogurt intake twice daily with or without added spices with a two-week washout period between study arms.
Who Masked: Investigator
Masking Description: The study coordinator and participants are unblinded due to the nature of the study design and intervention; however, the PI will remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm - Yogurt with added Spices (Experimental): Consumption of twice daily yogurt with added spices for four weeks.
  Interventions: Other: Yogurt with added Spices
- Sham Arm - Yogurt without added Spices (Sham Comparator): Consumption of twice daily yogurt without added spices for four weeks.
  Interventions: Other: Yogurt without added Spices

INTERVENTIONS:
Other: Yogurt with added Spices — Consumption of twice daily yogurt with added spices for four weeks.
  Arms: Intervention Arm - Yogurt with added Spices
Other: Yogurt without added Spices — Consumption of twice daily yogurt without added spices for four weeks.
  Arms: Sham Arm - Yogurt without added Spices

SUMMARY:
Among food products receiving attention for prebiotic functionality, spices represent a flavorful vehicle for cultivating a healthy gut microbiota. As the required doses of spice-derived polyphenols to elicit prebiotic and systemic metabolic effects are not well-characterized, additional research is warranted. Thus, the investigators propose to use a food-first synbiotic (prebiotic + probiotic) approach to examine alterations in the gut microbiota pre- and post-intervention/placebo and their relationship with systemic cardiometabolic effects mediated by short chain fatty acids (SCFA) and gut-derived metabolites.

DETAILED DESCRIPTION:
Study will be conducted as a single blind, randomized crossover design with a 4-week arm (placebo or control) followed by a 2-week washout period and another 4-week arm (placebo or control).

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women ages 50-69y with a BMI of 18.5 - 34.9 kg/m2

Exclusion Criteria:

* Dx - Diagnosis of cardiovascular disease, type 1 or 2 diabetes, liver disease, cancer, endocrine disorders, or inflammatory condition such as rheumatoid arthritis.
* GI - History of gastrointestinal surgery, irritable bowel syndrome, intestinal bowel disease, or other gastrointestinal distress such as chronic diarrhea, bulimia, anorexia, or frequent laxative use
* Rx or Supplements - Actively taking steroids or antibiotics in the previous two to three months, or currently using tobacco products, > 10% weight loss or gain in the last 6 months, unwilling to stop taking prebiotic/probiotic or fiber supplements
* Dietary - Adherence to a high fiber/polyphenol rich diet, have an allergy, aversion, or intolerance to food and spices provided in this study

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Concentration of fecal short chain fatty acids including acetate, proprionate, and butyrate | pre/post each four-week study arm
  Units - uM
Concentration of serum leptin | pre/post each four-week study arm
  Units - ng/mL
Concentration of serum ghrelin (pg/mL) | pre/post each four-week study arm
  Units - pg/mL
Concentration of serum peptide tyrosine tyrosine (PYY) | pre/post each four-week study arm
  Units - pg/mL

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Alabama, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No